CLINICAL TRIAL: NCT04418596
Title: Integrated Longitudinal Research on the Etiology of CAM Deformity in Adolescent Male Elite Soccer Players and Matched Control
Brief Title: Longitudinal Follow-up of Male Soccer Players Prone to Developing CAM Hip Deformity
Acronym: CAM-FAI
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Other Study IDs: S62916
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Femoro Acetabular Impingement; CAM
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elite Soccer Players: Adolescent male aged 12-16 years old elite athletes that are recruited from special sport school in Leuven-Belgium and play football at a high level.
  Interventions: Radiation: bi-planer radiography (EOS), Conventional radiography (Hip+pelvis)
- Recreational Soccer players (control): Adolescent male aged 12-16 years old recruited from ordinary school in Flanders Belgium that play soccer or any other sport recreationally with no high intensity training
  Interventions: Radiation: bi-planer radiography (EOS), Conventional radiography (Hip+pelvis)

INTERVENTIONS:
Radiation: bi-planer radiography (EOS), Conventional radiography (Hip+pelvis) — low dose radiation medical imaging to visualise the hip joint and lumbo-pelvic complex specifically.
  Other Names: Clinical Screening; Motion Analysis

SUMMARY:
Femoroacetabular impingement (FAI) is a clinical problem in which abnormal contact occurs between the thighbone and the hip socket. In intensive, mostly still young, male athletes, this problem seems to be related to a bony deformity on the head of this thighbone, a so-called CAM. FAI itself gives rise to pain symptoms, but in time can even lead to premature osteoarthritis. However, the cause of a CAM deformity itself, nor how FAI then arises, is insufficiently known. In view of FAI prevention and its better treatment, this project thus tries to better understand the underlying mechanisms. For this purpose, we will combine detailed biomechanical evaluations of specific movement patterns with advanced medical imaging and state of the art clinical evaluations to longitudinally follow up a group with a known high risk of developing a CAM deformity, being young male elite soccer players. Findings within this study will be additionally compared with similar analyses performed in patients with FAI. This research aims to thus form a basis to define novel (sports-specific) training schemes for the prevention of FAI, but also to define the actual treatment and rehabilitation plans in more patient-specific and a better-informed way.

DETAILED DESCRIPTION:
This is a longitudinal follow-up study in which subjects are invited for data collection twice, the baseline time-point and the two years time-point.

Population:

12-16 years old male soccer players (40 elite level players , and 40 recreational level players)

In both data collection time-points the following measurements are preformed:

1. Clinical screening of hip joint
2. Radial MRI of bilateral hips
3. Biplanar and conventional x-ray Imaging of hip and pelvic region
4. Athlete-specific 3D motion analysis
5. Questionnaires on injury history and physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* For the the Elite Group: Playing soccer at high level and training for more that 10 hours a week
* For the Control group: Playing soccer or any other sport recreationally for a less than 5 hours a week

Exclusion Criteria:

* No prior history of major trauma or injury to the lower limbs and spine
* No prior history of neurological conditions that can effect movement and mobility

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Genetic component of being a male is required .
Study Population: Adolescent healthy males that are starting the final age of skeletal maturity(12-18 years of age). The 2 groups of the study are separated principally on the frequency and intensity of their athletic training.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The formation of CAM deformity on the anterior head-neck junction of the femur | two years post baseline measurements
  Detected using alpha angle on MRI/ Dunn's View x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Ghijselings, M.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University of Leuven Hospitals, Leuven, Flanders, Belgium